CLINICAL TRIAL: NCT00660725
Title: An Open Label Phase I Study of Gemcitabine/Oxaliplatin (GEMOX) and Vandetanib (ZACTIMA; ZD6474) Combination in Patients With Advanced Solid Malignancy (IRUSZACT0070) (UPCI 07-025)
Brief Title: Study of GemOx and Vandetanib in Advanced Solid Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leonard Appleman (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Leonard Appleman, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-025; IRUSZACT0070; UPCI 07-025
Record Dates: First submitted 2008-04-08; First posted 2008-04-17 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Incurable Solid Malignancy
Keywords: Gemcitabine; Oxaliplatin; Vandetanib; Phase I
MeSH Terms: interventions — vandetanib; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib/GEMOX (Other): All subjects receive the same combination study drug and follow the same study schedule. As a phase 1 study, only the doses will vary between subjects.
  Interventions: Drug: Vandetanib; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Vandetanib — Vandetanib is a pill that will be self-administered orally on Days 1-14 of each 14-day cycle. The dose of vandetanib each subject will receive will be determined by a dose escalation schedule (either 200 mg or 300 mg per day), which will be followed to determine the MTD of the study drug combination (vandetanib + GemOx). In the absence of disease progression, unacceptable toxicities, or other complications, the vandetanib and GemOx combination may continue per protocol for a maximum of 6 cycles, or 12 weeks. In subjects who show response or stable disease, vandetanib may be continued as a single agent beyond the 6 cycle maximum, at the investigator's discretion.
  Other Names: Zactima; ZD6474
Drug: Gemcitabine — 30-minute IV infusion of 1000 mg/m^2 gemcitabine on Day 1 of each 14-day cycle.
  Other Names: Gemzar®
Drug: Oxaliplatin — Immediately following gemcitabine IV: 2-hour IV infusion of 85 mg/m^2 oxaliplatin on Day 1 of each 14-day cycle.
  Other Names: Eloxatin®

SUMMARY:
This is a research study that will try to find the highest and safest dose of an experimental drug, vandetanib, that can be given in combination with two standard chemotherapy agents, gemcitabine and oxaliplatin, to subjects with advanced solid malignancies.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalating, non-randomized study of the safety and tolerability of vandetanib in combination with a fixed dose of gemcitabine and oxaliplatin (GemOx) in the treatment of patients with advanced solid malignancy. EGFR is an important target for therapeutic drug development. It is widely expressed in most cancers and has a vital role in the regulation of proliferation signals. EGFR is expressed in a high degree (>80%) of pancreatic tumors and is a rational target for therapy. Vandetanib selectively inhibits EGFR tyrosine kinase activity and VEGF-2 receptor. It has good oral bioavailability and has growth inhibitory activity in a wide variety of human cell lines including cells with acquired resistance to other EGFR inhibitors. The growth inhibitory property of vandetanib in vivo correlates more with its anti VEGF property, especially in cell lines with acquired resistance to EGFR inhibition. The combination of gemcitabine and oxaliplatin (GEMOX) is a well-established regimen that has demonstrated encouraging antitumor activity in pancreaticobiliary cancers in phase II studies. Recent clinical trials have also shown activity in hepatobiliary and germ cell tumors. The combination of vandetanib and gemcitabine has potential advantages and may result in an additive or synergistic effect. The GEMOX regimen is well tolerated, and toxicity does not overlap with the most common toxicity of rash or diarrhea observed with vandetanib. Thus, the combination of vandetanib and GEMOX is expected to be a well tolerated, and an easily administered regimen with improved efficacy and no overlapping toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced incurable solid malignancy who are likely to benefit from GEMOX therapy.
* Provision of informed consent prior to any study procedures.
* Females and males age ≥18 years
* Histological/cytological confirmation of malignancy
* Negative pregnancy test for women of childbearing potential
* ECOG performance status of 0 or 1
* Ability to take oral medications without difficulty
* Adequate bone marrow function: ANC >1500/L and platelet count >100,000/dL
* Adequate hepatic function: Total Bilirubin ≤ 1.5 x ULN, ALT/AST ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis), ALP ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis)
* Serum calcium in normal range (ionized or adjusted for albumin), Serum magnesium in normal range, Serum Potassium ≥ 4.0 mmol/L. Supplementation allowed.
* Serum Cr < 1.5 x UNL or Creatinine Clearance ≥ 50 mL/min calculated by Cockcroft-Gault formula
* Men and women of childbearing potential must be willing to practice acceptable methods of birth control.
* Patients with brain metastasis should have received appropriate therapy and have stable disease at least 4 weeks after radiotherapy/surgery.
* Subjects should have recovered from side effects of prior therapy to grade 1 or less

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of QTc prolongation with other medications that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block (LBBB.)
* QTc with Bazett's correction that is unmeasurable, or ≥480 msec on screening ECG. (Note: If a subject has a QTc interval ≥480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the subject to be eligible for the study.) Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is ≥ 460 msec.
* Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes.
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Currently active diarrhea that may affect the ability of the patient to absorb the vandetanib or tolerate diarrhea.
* Women who are currently pregnant or breast feeding.
* Receipt of any investigational agents within 30 days or commercially available agents within 21 days prior to commencing study treatment
* Last dose of prior chemotherapy discontinued less than 4 weeks before the start of study therapy
* Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy for less than 12 fractions
* Any unresolved toxicity greater than CTCAE grade 1 from previous anti-cancer therapy
* Previous enrollment or randomization of treatment in the present study
* Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy
* Peripheral neuropathy grade 2 or of greater severity of any cause
* More than 2 prior systemic chemotherapy regimens for advanced stage disease. Prior adjuvant chemotherapy will not count as a prior regimen.
* Known severe hypersensitivity to vandetanib or any of the excipients of these products.
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
* Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of CYP3A4 function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To establish the Maximum Tolerated Dose (MTD) and toxicities of vandetanib (Zactima; ZD6474) in combination with fixed dose of GEMOX (gemcitabine/oxaliplatin) and to establish the recommended phase II dose of the GEMOX and vandetanib regimen | The MTD (and recommended phase II dose) is defined as the highest dose at which <2 of 6 patients experience DLT. The observation period for DLT is the first cycle of therapy.

SECONDARY OUTCOMES:
To document clinical responses and to identify time to progression (TTP) of each patient compared to TTP on prior therapy | Radiologic imaging is done every 6-7 weeks for disease assessment

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J. Appleman, M.D., Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute / Hillman Cancer Center, Pittsburgh, Pennsylvania, United States